CLINICAL TRIAL: NCT03409393
Title: Feasibility and Relevance of High-Intensity Functional Training in Patients Undergoing Specialised Early Intervention Treatment for First-Episode Psychosis
Brief Title: Feasibility and Relevance of High-Intensity Functional Training in Patients With First-Episode Psychosis
Acronym: COPUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University of Copenhagen (Other); Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Responsible Party: Principal Investigator, Julie Midtgaard, Associate Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: COPUS; 119481 (Other Grant/Funding Number: TrygFonden)
Record Dates: First submitted 2018-01-04; First posted 2018-01-24 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Schizophrenia; Schizotypal Disorder; First Episode Psychosis; Psychotic Disorders; Schizoaffective Disorder
Keywords: Human; Denmark; Adult; Adolescent; Young Adult; Male; Female; Physical Activity; Maximum Oxygen Consumption; Resistance Training; High-Intensity Functional Training; Aerobic Exercise; Motivation; Feasibility; Relevance; Health Behavior
MeSH Terms: conditions — Schizophrenia; Schizotypal Personality Disorder; Psychotic Disorders; Motor Activity; Health Behavior

STUDY DESIGN:
Intervention Model Description: The participants will be randomly assigned (1:1) to either an Intervention Group that in the initial study phase (week 0-8) receives the COPUS intervention plus usual care (i.e. OPUS treatment) or to a Control Group that only receives usual care in the initial phase. In the second phase of the study (week 8-16), participants allocated to the control group are offered the COPUS intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The COPUS intervention plus usual care (OPUS treatment).
  Interventions: Other: The COPUS intervention; Other: Usual Care (OPUS treatment)
- Control Group (Other): Usual care (OPUS treatment).
  Interventions: Other: Usual Care (OPUS treatment)

INTERVENTIONS:
Other: The COPUS intervention — The COPUS intervention consists of 8 weeks of High-Intensity Functional Training (HIFT). The frequency of the training is 3 sessions per week and the duration is one hour per session. The intervention is group-based and supervised. Each training session includes warm-up (15 min), followed by 30 minutes of HIFT based on a range of varied functional exercises, including elements of strength training and aerobic exercise. The sessions are supervised by a trained physiotherapist and exercise physiologist supported by 2 two trained bachelor students in Sports Science.
  Arms: Intervention Group
Other: Usual Care (OPUS treatment) — Usual care include specialised early intervention treatment (OPUS treatment) and consists of three main pillars: modified assertive treatment, family involvement, and social skill training. OPUS treatment is delivered via multidisciplinary teams include psychiatrists, psychologists, nurses, social workers, physiotherapists, and vocational therapists. All team members, except for the psychiatrist, function as case managers. The ratio of patients to case managers must not exceed 12:1.

SUMMARY:
The aim of the COPUS study is to investigate, whether it is possible to recruit and retain young people with first-episode psychosis, to an 8 week supervised High-Intensity Functional Training intervention (HIFT) (i.e. COPUS Intervention) and to investigate if oxygen uptake, body composition and physical function improves following participation in the intervention.

DETAILED DESCRIPTION:
The introduction of specialized early intervention (SEI) is stated to be the most successful recent addition to the treatment of schizophrenia and other psychotic illnesses. In Denmark, SEI teams called OPUS, offer early intervention treatment (i.e. OPUS treatment) to young patients between 18 and 35 years with first-episode psychosis. The OPUS treatment consists of three main pillars: modified assertive treatment, family involvement, and social skill training. OPUS treatment is delivered via multidisciplinary teams including psychiatrists, psychologists, nurses, social workers, physiotherapists, and vocational therapists.

Despite considerable progress in treatment of schizophrenia, people diagnosed with schizophrenia live significantly shorter lives, compared to the rest of the population. The higher mortality rate can be partly explained by an increased risk of cardiovascular disease, including metabolic syndrome, which may be documented already in the first months after start of medical anti-psychotic treatment. It is widely acknowledged that physical activity constitutes a cornerstone in the prevention of cardiovascular disease and metabolic syndrome. Therefore, despite the influence of non-modifiable factors (e.g. genetics), it is reasonable to assume that physical activity can promote health and prevent somatic disease in people diagnosed with schizophrenia.

However, currently, physical activity is not included in early intervention treatment of schizophrenia. Moreover, people with schizophrenia may experience anxiety, loss of motivation, apathy and social isolation, which can constitute significant barriers for adherence to physical activity. Existing knowledge in relation to physical activity behaviour change and adoption is therefore difficult to transfer directly to people with schizophrenia. Development and testing of new initiatives, which can be integrated into clinical practice, and offered complementary to SEI are thus warranted.

Against this background, the aim of the current study (called the COPUS study) is to investigate, whether it is possible to recruit and retain young people with first-episode psychosis, to an 8-weeks supervised High-Intensity Functional Training (HIFT) intervention (i.e. COPUS intervention) and to investigate if oxygen uptake, body composition and physical function changes following participation in the COPUS intervention. The study is organized as a randomized mixed methods feasibility study.

The COPUS intervention is offered in a private fitness centre in the local community. The intervention contains three training sessions of one hour duration per week, with the recommendation to the participants, to take part in at least two sessions per week.

The investigators aim to include 30 participants whom will be randomly assigned (1:1) to either an intervention group receiving the COPUS intervention plus usual care (i.e. standard OPUS treatment) or a control group including only receiving usual care (i.e. standard OPUS treatment). Participants allocated to the control group are offered the COPUS intervention after eight weeks.

The design and choice of methods reflect the complexity of the intervention (combination of social and physical elements that are difficult to control and isolate) and the desire to establish a scientifically informed basis for a subsequent, up-scaled, pragmatic randomized multicentre study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 35 years
* Diagnosed with Schizophrenia or Schizotypal disorders
* Undergoing OPUS treatment for at least 6 months or stabilized medical anti-psychotic treatment
* Danish speaking

Exclusion Criteria:

* Physical contraindications for physical activity
* Pregnant (self-reported)
* Unable to give adequately informed consent
* Mentally disabled

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Assessment of changes in Physical Fitness (VO2max) | Change from Baseline Physical Fitness (VO2max) at 2 months.
  Assessed by the maximum amount of oxygen the body can utilize during a specified period of intense exercise.
Recruitment Rate | Registration of recruitment occurs in the 4 weeks prior to the baseline tests.
  Registration of patients enrolled in the study compared to the total number of eligible patients.
Retention Rate | From baseline up to 4 months.
  Registration of the participants attendance in the High-Intensity Functional Training compared with the number of possible training sessions during the period.

SECONDARY OUTCOMES:
Assessment of changes in body weight | Change from Baseline Body Weight at 2 months.
  The participants are placed on a bioelectric impedance scale which is a non-invasive valid measurement method for determining body weight.
Assessment of changes in fat percentage | Change from Baseline Fat Percentage at 2 months.
  The participants are placed on a bioelectric impedance scale which is a non-invasive valid measurement method for determining fat percentage.
Assessment of changes in bone mass | Change from Baseline Bone Mass at 2 months.
  The participants are placed on a bioelectric impedance scale which is a non-invasive valid measurement method for determining bone mass.
Assessment of changes in muscle mass | Change from Baseline Muscle Mass at 2 months.
  The participants are placed on a bioelectric impedance scale which is a non-invasive valid measurement method for determining muscle mass.
Assessment of changes in Visceral Fat | Change from Baseline Visceral Fat at 2 months.
  The participants are placed on a bioelectric impedance scale which is a non-invasive valid measurement method for determining visceral fat.
Assessment of changes in Resting Blood Pressure | Change form Baseline Resting Blood Pressure at 2 months.
  The participants' Resting Blood Pressure are tested according to the American Heart Association practice guidelines for blood pressure Measurement.
Assessment of changes in countermovement jump height | Change form Baseline Jump Height at 2 months.
  Determination of potential changes in countermovement jump height measured using the non-invasive Optojump system (www.optojump.com)
Assessment of changes in Leg Muscle Strength | Change form Baseline Leg Muscle Strength at 2 months.
  Determination of potential changes in leg muscle strength by the non-invasive 30-Second Chair Stand test. The test measures how many times the participant can reach a full standing position from a sitting position in 30 seconds. Score range from 0 and up with a higher score being considered as a better outcome.
Assessment of changes in Hand Grip Strength | Change form Baseline Hand Grip Strength at 2 months.
  Determination of potential changes in grip strength measured quantitatively using a hand dynamometer.
Assessment of changes in Balance | Change form Baseline balance at 2 months.
  Determination of potential changes in balance using the Flamingo Balance Test. The participant stands on a 3 centimeter wide beam while holding the instructors hand. The tests then measures how many times the participant loses balance in 60 seconds.Score range from 0 and up with a lower score being considered as a better outcome.
Assessment of changes in Self-reported Physical Activity Behavior | Change from Baseline Physical Activity Behaviour at 2 months.
  Assesment of changes in self-reported physical activity behaviour using the Physical Activity Scale (PAS). The PAS measures self-reported amount of time spent on different physical activities, such as sports, work, and leisure time during 24 hours on an average weekday. The activities are organized in nine different metabolic equivalent (MET) levels ranging from sleep/rest (0.9 METs) to high-intensity physical activities (>6 METs). MET is the Metabolic Equivalent of Task and is a physiological measure expressing the energy cost of physical activities and is defined as the ratio of metabolic rate (and therefore the rate of energy consumption) during a specific physical activity to a reference metabolic rate. Therefore, higher MET scores in the Physical Activity Scale indicates a better outcome than lower scores.

OTHER OUTCOMES:
Monitoring of training intensity (for the Intervention Group only) | Through study completion, an average of 4 months
  Determination of whether the training intensity is adequate to increase Physical Fitness, the workload during training is continuously measured. A validated device called Actiheart which is both an accelerometer and a heart rate monitor is used to measure workload.
Adverse events | Through study completion, an average of 4 months
  We will continuously record adverse events that may arise as a result of the intervention, including physical damage, discomfort and any deterioration of symptoms. The adverse events will be registred both in the intervention period and in the Control Group training period.
Resource Consumption | Through study completion, an average of 4 months
  In order to evaluate the sustainability of the intervention, we want to register how much time (in minutes) OPUS staff spends on the project

CONTACTS AND LOCATIONS:
Overall Officials: Julie Midtgaard, Ph.D., Principal Investigator — The University Hospitals Centre for Health Research (UCSF) / Copenhagen University Hospital (Rigshospitalet); Helle Schnor, Ph.D., Study Director — Mental health services in the Capital Region of Denmark, Psychiatric Center Glostrup
Locations (1):
- OPUS, Brøndby, Denmark

REFERENCES:
- [Derived] Midtgaard J, Schnor H, Bjerre ED, Jespersen T, Jelsoe N, Frolund N, Seier S, Ronbog JW, Nordsborg NB, Ebdrup BH. Exercise training complementary to specialised early intervention in patients with first-episode psychosis: a feasibility randomised trial. Pilot Feasibility Stud. 2021 Aug 19;7(1):162. doi: 10.1186/s40814-021-00900-5. PMID 34412705
- [Derived] Larsen LQ, Schnor H, Tersbol BP, Ebdrup BH, Nordsborg NB, Midtgaard J. The impact of exercise training complementary to early intervention in patients with first-episode psychosis: a qualitative sub-study from a randomized controlled feasibility trial. BMC Psychiatry. 2019 Jun 21;19(1):192. doi: 10.1186/s12888-019-2179-3. PMID 31226959
- See also: Official institutional website — http://www.ucsf.dk